CLINICAL TRIAL: NCT03803397
Title: A Study to Evaluate the Safety and Efficacy of Intratumoral Injection of PV-001-DV in Combination With Infusion of PV-001-DC in Patients With Advanced Melanoma
Brief Title: Arm 1: Lysate Pulsed Dendritic Cells (PV-001-DC) in Patients With Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PrimeVax Immuno-Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV001-001 (Arm 1)
Record Dates: First submitted 2018-12-31; First posted 2019-01-14 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PV-001-DC alone (Experimental): Autologous Monocyte-derived Lysate Pulsed Dendritic Cells
  Interventions: Biological: PV-001-DC

INTERVENTIONS:
Biological: PV-001-DC — Patient-specific cellular therapeutic for cancer immunotherapy

SUMMARY:
Autologous monocyte-derived dendritic cells pulsed with tumor lysate (PV-001-DC) will be given to a group of 3 people. If this is found to be safe, it will be given to up to 7 other people, for a total of up to 10 people in this arm. This will be the first study of PV-001-DC.

Eligible patients must be progressing after having completed prior therapy with a PD-1/PD-L1 antagonist alone or in combination with anti-CTLA-4. If the patient is positive for BRAF, the patient must have progressed on at least one BRAF inhibitor in addition to a PD-1/PD-L1 inhibitor alone or in combination with CTLA-4 for metastatic melanoma.

Although other kinds of dendritic cells (DCs) have been approved to treat some forms of cancer, they have not been approved to treat melanoma. PV-001-DC is a special kind of DCs that is combined with tumor lysate. The study procedures will start with the removal of a small amount of tumor tissue processed into protein fragments (lysate). There will also be collection of white blood cells through apheresis (a procedure in which blood is drawn from a patient and separated into its different cell types), the white blood cells will be collected and the remainder returned to the patient. Dendritic cells will be grown from the collected white blood cells and combined with the lysate to form PV-001-DC.

On the first day of study treatment, patients will go to the clinic and have a needle placed in a vein. The PV-001-DC product will be infused into the patient's vein. Approximately every 3 weeks, for a total of 4 treatments, patients will receive additional infusions of PV-001-DC. Patients will be at the clinic for at least 1 hour following the end of the PV-001-DC infusion and if they feel fine, they may go home.

Scans will be performed during the study at different times to see if their tumors have changed in size. Patients will also have their blood and small samples of tumors tested for changes to the immune system. After 365 days, the trial will be completed for that patient.

Investigators will monitor patients carefully for any harmful side effects. The side effects in people cannot be completely known ahead of time

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed patients with un-resectable AJCC Stage III or IV melanoma who have measurable disease. Measurable disease is required, and is defined as tumor can be measured in two dimensions.
* Patient must have progressed with prior therapy with a PD-1 / PD-L1 antagonist alone or in combination with anti-CTLA-4. If the patient is positive for BRAF, the patient must have progressed on at least one BRAF inhibitor in addition to a PD-1 / PD-L1 inhibitor alone or in combination with CTLA4 for metastatic melanoma.
* Tumor specimens must be available for tumor lysates and immunological studies.
* ECOG Performance Status of ≤ 2 (corresponds to a Karnofsky Performance Status (KPS) of ≥ 70).
* Patients must be 18 years or older and able to give informed consent.
* Adequate bone marrow function of White Blood Cell (WBC) count to ≥ 1,500/uL; platelet count ≥ 100,000/mm3; absolute neutrophil count (ANC) > 1,200/uL
* Patients must have adequate renal function by serum creatinine of ≤ 2.0 mg/dL.
* Adequate hepatic function of bilirubin ≤ 2.5 mg/dL; SGOT/SGPT < 3× upper limit of normal (ULN).
* Patients must have the required wash out periods from prior therapy:

  * Topical therapy: 2 weeks.
  * Chemotherapy and radiotherapy: 4 weeks.
  * Other investigational therapy: 4 weeks
* Patients of reproductive potential and their partners must agree to use an effective (>90% reliability) form of contraception during the study and for 4 weeks following the last study drug.
* Women of reproductive potential must have a negative urine pregnancy test.
* Patients should have a life expectancy of > 6 months.
* Patient should be able to comply with the treatment schedule and have the ability to understand and willingness to sign the informed consent document.
* Patients with manageable central nervous system metastases may be selected to this trial. The CNS metastases are defined as manageable if there is no progression for at least 4 weeks as determined by clinical examination and brain imaging (MRI and/or CT).

Exclusion Criteria:

* Pre-existing autoimmune or antibody mediated disease including systemic lupus erythematous, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
* Known history of human immunodeficiency virus (HIV) or any active immunosuppressive systemic infection or a suppressed immune system, including acquired immuno-deficiency syndrome (AIDS) or HIV positivity and known hepatitis infections (HCV or HBC), as assessed by serology.
* Patients on immunosuppressive therapy. Concurrent steroid use of not more than an equivalent of 10 mg of prednisone is allowed.
* Previous organ transplantation.
* Patients with active infection or with a fever >101°F (38.5°C) within 3 days prior to the first scheduled treatment.
* Concurrent participation in other treatment related clinical studies. Non-treatment studies (e.g. observation or tumor cell analysis studies) are allowed.
* Prior malignancy (active within 3 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.

  o Significant cardiovascular disease (i.e., New York Heart Association (NYHA) class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
* Female patients who are pregnant or lactating.
* Patients taken off Checkpoint Blockade agents: Ipilimumab, Nivolumab, Pembrolizumab, for Grade 3 or greater autoimmune toxicity.
* Patients who are positive for B-RafV600 mutation and are responding to targeted therapy.
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with his/her participation in the study, or to interfere with the interpretation of the results.
* Patients with endocrinopathy greater than grade III.
* Patients who have undergone a splenectomy in their previous medical history will be excluded from this trial. Evidence of a splenectomy will be from history or records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events | 365 days
  Treatment-Emergent Adverse Event Incidence in patients receiving IV infusion of PV-001-DC

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 365 days
  Tumor response will be measured per investigator's assessment according to RECIST v1.1 and iRECIST
Progression-Free Survival (PFS) | 365 days
  The length of time during the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse, up to the end of the study
Overall Survival (OS) | 365 days
  Overall Survival is measured from the date of enrollment to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date, up to the end of the study

IPD SHARING:
Plan to Share IPD: No